CLINICAL TRIAL: NCT00003633
Title: Treatment of Prostate Cancer by Induction of Alternate Cell Death Pathways: A Phase I Trial of Docetaxel, Estramustine, Mitoxantrone and Prednisone
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066717; CPMC-IRB-8040; CPMC-IRB-8040-2/9173; NCI-V98-1487; CPMC-IRB-AAAA5741
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2005-03

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; Mitoxantrone; Prednisone

INTERVENTIONS:
Drug: docetaxel
Drug: estramustine phosphate sodium
Drug: mitoxantrone hydrochloride
Drug: prednisone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of combination chemotherapy in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated doses of docetaxel and mitoxantrone in combination with a fixed dose of estramustine and prednisone, when given to patients with advanced prostate cancer.
* Characterize the toxicity of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of mitoxantrone and docetaxel. Patients are stratified into one of two risk groups (good risk group or poor risk group) based on the number of prior chemotherapy regimen(s) and the occurrence and sites(s) of prior radiation.

All patients receive oral prednisone twice daily on days 0-3, oral estramustine three times daily on days 1-5, mitoxantrone IV bolus on day 2, and docetaxel IV over 1 hour on day 2. Courses repeat every 21 days in the absence of unacceptable toxicity and disease progression. Patients with stable disease may go off treatment after 6 courses.

Dose escalation proceeds independently for each risk group. Cohorts of 3 patients are entered into each risk group. If 1 of 3 patients at a dose level experiences dose limiting toxicity (DLT), then 3 additional patients are accrued into this level. If 2 of 6 patients at a dose level experience DLT, then dose escalation stops and the maximum tolerated dose (MTD) is defined at the previous dose level. At least 6 patients must be treated at the MTD.

Patients are followed every 3 months until death.

PROJECTED ACCRUAL: At least 12 patients (6 in each risk group) will be accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Failure of complete androgen ablation (orchiectomy or LHRH and antiandrogen therapy) as manifested by at least 1 of the following criteria:

  * Rise in serum PSA greater than 50% of nadir confirmed on 2 measurements 1 week apart
  * Appearance of new lesions on bone scan
  * Appearance of new soft-tissue lesions
* Measurable or evaluable disease
* No brain or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 3 months

Hematopoietic:

* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* SGOT and SGPT no greater than 2 times ULN

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No history of coagulopathy
* No myocardial infarction in the last 6 months
* No history of cardiovascular accident
* No history of congestive heart failure

Neurological:

* No symptomatic peripheral neuropathy greater than grade 1
* No history of significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures

Pulmonary:

* No history of pulmonary embolus

Other:

* Testosterone no greater than 3.5 nmol/L
* No contraindications to glucocorticoid therapy such as uncontrolled diabetes mellitus or active peptic ulcer disease
* No active infection
* No other serious illness or medical condition
* No other concurrent or prior malignancy in the past 5 years except previously excised or curatively irradiated nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hormonal therapy (including nonsteroidal antiandrogens, but not LHRH agonists)

Radiotherapy:

* No prior radiotherapy to greater than 30% of bone marrow
* At least 6 weeks since isotope therapy
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since prior investigational drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P. Petrylak, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States